CLINICAL TRIAL: NCT01515644
Title: A Randomized, Double-blind, Controlled Study on the Effect of Inulin on Gut Health of Infants
Brief Title: Study on the Effect of Inulin in Infant Formula on Gut Health
Acronym: STAR-IFFO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: PT. Sari Husada (Industry)
Collaborators: Danone Global Research & Innovation Center (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CT.01.2010
Record Dates: First submitted 2012-01-05; First posted 2012-01-24 (Estimated); Last update posted 2013-04-24 (Estimated); Status verified 2013-04

CONDITIONS: Healthy Infants
Keywords: Healthy infants; Infant formula; Prebiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Intervention group I (Experimental): Intervention group I: Powder based Infant formula with Inulin I
  Interventions: Other: Powder based infant formula
- Intervention group II (Experimental): Intervention group II: Powder based Infant formula with Inulin II
  Interventions: Other: Powder based infant formula
- Intervention group III (Placebo Comparator): Intervention group III: Powder based Infant formula without Inulin
  Interventions: Other: Powder based infant formula

INTERVENTIONS:
Other: Powder based infant formula — Powder based infant formula with Inulin I
  Arms: Intervention group I
Other: Powder based infant formula — Powder based infant formula with Inulin II
  Arms: Intervention group II
Other: Powder based infant formula — Powder based infant formula without Inulin
  Arms: Intervention group III

SUMMARY:
In this study the effect of Infant formula with added Inulin will be compared with the effect of Infant formula without Inulin on the Bifidobacterium level in stool.

It is expected that drinking Infant formula with added Inulin will result in higher beneficial bacteria level in stool compared to an Infant formula without Inulin.

ELIGIBILITY:
Inclusion criteria at screening:

* Healthy infants between 3-4 months (91-120 days after birth) of age at day 1 of the study, with healthy growth determined based on WHO standard
* Fully formula-fed in the 28 days prior to inclusion
* Expected investigational product intake of min 500ml per day
* Written informed consent from the parents

Exclusion criteria at screening:

* Low birth weight (LBW) less than 2,000g.
* Disorders requiring a special diet (such as food intolerance or food allergy or complaints such as reflux, constipation and cramps for which special toddler formula is required)
* Use of systemic antibiotics or antimycotics medication in the 14 days prior to the study
* Significant congenital abnormality that will interfere with the study objectives in the opinion of the investigator.
* Investigator's uncertainty about the willingness or ability of the parents to comply with the protocol requirements.
* Participation in any other studies involving investigational or marketed products concomitantly or within two weeks prior to entry into the study.

Exclusion criteria for intervention period:

* Not consuming study product longer than 2 days consecutively
* Intake of study product is less than 500ml per day for 7 days

Ages: 3 Months to 4 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 164 (Actual)
Dates: Start 2011-10; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Difference between beneficial bacteria I level in stool at week 4 and week 8. | Week 4, Week 8.

SECONDARY OUTCOMES:
Difference between beneficial bacteria II level in stool at week 4 and week 8. | Week 4, Week 8.
Difference between pH of stool at week 4 and week 8. | Week 4, Week 8.
Difference between stool consistency at week 4 and week 8. | Week 4, Week 8.
Difference between sIgA at week 4 and week 8. | Week 4, Week 8.
Difference between SCFA at week 4 and week 8. | Week 4, Week 8.
Safety and tolerability. | From date of baseline visit (day 1) until the date of visit 8 (day 56)
  The safety and tolerability achieved by continuous recording of adverse events, including the occurrence of diarrhea and constipation.

CONTACTS AND LOCATIONS:
Overall Officials: Hanifah Oswari, dr., Sp.A(K), PhD, Principal Investigator — Research Unit of Indonesian Pediatrics Association
Locations (1):
- Research Unit of Indonesian Pediatrics Association, Jakarta, Indonesia